CLINICAL TRIAL: NCT06021405
Title: A Prospective Study to Investigate the Pathophysiology of the Koebner's Phenomenon in Psoriasis and Lichen Planus
Brief Title: Koebner's Phenomenon in Psoriasis and Lichen Planus
Acronym: RENBOEK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marie-Charlotte Brüggen (Other)
Responsible Party: Sponsor-Investigator, Marie-Charlotte Brüggen, Prof. Dr. med. PhD, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-00427
Record Dates: First submitted 2023-08-11; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Kobner Phenomenon; Psoriasis; Lichen Planus
MeSH Terms: conditions — Psoriasis; Lichen Planus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tape stripping (Experimental)
  Interventions: Procedure: Tape stripping

INTERVENTIONS:
Procedure: Tape stripping — a small area of skin will be tape-stripped with adhesive tape for up to 40 times and/or rubbed with a wooden spatula until the skin shows a slight erythema

SUMMARY:
Psoriasis and lichen planus often occur at mechanically irritated skin sites (e.g. tight clothing). The investigators would like to investigate this phenomenon in more detail in this study. For this purpose, the skin is specifically irritated at a small and cosmetically favorable site by tearing off scotch tape or rubbing with a wooden spatula. In order to be able to examine the inflammatory processes caused by the irritation more closely, a small skin sample and a skin swab are taken from the irritated area. This skin sample and the swab are repeated after three and fourteen days.

ELIGIBILITY:
Inclusion Criteria:

* Dermatologist diagnosed psoriasis (group psoriasis), lichen planus (group lichen planus) or no skin disease (group healthy controls)
* Subject is capable of giving informed consent
* Signed informed consent

Exclusion Criteria:

* Use of systemic immunosuppressive/immunmodulating agents in the last three months
* Use of topical anti-inflammatory treatment in the last 7 days in the area of sampling.
* Phototherapy in the last 4 weeks
* Active or recurrent serious bacterial, fungal or viral infection at the time of enrollment by patient history, including patients with Human Immunodeficiency Virus (HIV) infection, Hepatitis B and Hepatitis C infection, active or untreated latent tuberculosis.
* Female patients of childbearing potential who are pregnant or breast feeding or planning a pregnancy during the duration of the trial and/or not practicing acceptable birth control for the duration of the trial
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2024-12-24 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Differences in the transcriptomic profile comparing psoriasis patients with and without induced koebner phenomenon | Day 0, Day 3 (optional), Day 14 (optional)
  Transcriptomic profile at all timepoints (reads per 55µm diameter dot)

SECONDARY OUTCOMES:
Differences in the proteomic profile comparing psoriasis patients with and without induced koebner phenomenon | Day 0, Day 3 (optional), Day 14 (optional)
  Olink multiplex proteomics analysis at all timepoints
Characterization of involved immune cells in the skin comparing psoriasis patients with and without induced koebner phenomenon | Day 0, Day 3 (optional), Day 14 (optional)
  Imaging mass cytometry (skin biopsies) at all timepoints
Characterization of skin mikrobiome | Day 0, Day 3, Day 14
  Skin swabs at all timepoints, analyzed by isolation and sequencing of the microbial DNA

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Charlotte Brüggen, MD PhD, Principal Investigator — University of Zurich